CLINICAL TRIAL: NCT01672658
Title: Standard Vestibular Rehabilitation Training (VRT) vs. Sensory Kinetics Balance System (SKBS) + VRT on Balance and Functional Outcomes in the Mild Traumatic Brain Injury (mTBI) Population.
Brief Title: Traditional Balance vs Vibrotactile Feedback Training for Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Edward Hines Jr. VA Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Arun Jayaraman, Research Scientist, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUSTU58913
Record Dates: First submitted 2012-08-14; First posted 2012-08-27 (Estimated); Results first posted 2016-04-04 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Traumatic Brain Injury; Vestibular Deficits
Keywords: TBI,; vestibular
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sensory Kinectics Balance System (Experimental): Subjects will be randomized in to one of two groups. The group that will receive training on the SKBS device along with traditional vestibular and balance training.
  Interventions: Device: Sensory Kinetics Balance System
- Traditional Vestibular Rehabilitation (Active Comparator): Traditional vestibular rehabilitation will include VOT exercises that will work toward increasing the gain of the system as well as walking, balance re-training, and functional mobility.
  Interventions: Other: Traditional Vestibular Rehabilitation

INTERVENTIONS:
Device: Sensory Kinetics Balance System — Subjects will participate in balance/gait/functional mobility training twice a week for 8 weeks.
  Arms: Sensory Kinectics Balance System
Other: Traditional Vestibular Rehabilitation — Subjects will perform traditional vestibular/balance rehabilitation which will include gait training, balance retraining, vestibular retraining, and functional mobility.
  Arms: Traditional Vestibular Rehabilitation

SUMMARY:
The goal of this clinical research study at RIC is to determine the value and benefit of the SK multimodal balance training system through independent clinical evaluations. The functional benefit of the SK Balance system will be measured by any improvements in balance and functional assessments.

This study is primarily funded through Engineering Acoustics as a subcontract for a phase II Small Business Innovation Research by the Department of Defense.

3) Hypotheses & Research Objectives and Purpose:

The specific research questions to be addressed are:

1. How does an 8-week SKBS+VRT training intervention compare to an 8-week standard VRT intervention on balance and functional gait measures in mild traumatic brain injury (mTBI) participants.
2. How do SKBS measurement tools compare to standard clinical assessments of gait and balance in mTBI patients The purpose of this clinical research study is to compare the value and benefit of the SK multimodal balance training system in combination with traditional vestibular rehabilitation vs. traditional vestibular rehabilitation alone through independent clinical evaluations. The functional benefit of the SK Balance system will be measured by any improvements in clinical measures of balance, functional mobility, and gait assessment.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) occurs when physical trauma causes temporary or permanent neurological damage. In some cases, symptoms can continue over time and contribute to disability. Dizziness and vertigo are associated with nearly all reported studies of mild Traumatic Brain Injury (mTBI) and are a significant and functionally limiting component of the overall disability.

TBI is one of the many risks faced by military personnel in combat activities . In a RAND Corporation survey of service members who had been deployed to Iraq or Afghanistan, 19% reported probable TBI. Dizziness and vertigo are associated with nearly all reported studies of mTBI and are a significant and debilitating component of the overall disability. mTBI are currently caused by both blast and impact injuries resulting in variable disabilities . Overt symptoms may include balance and spatial disorientation problems (vertigo) related to vestibular dysfunction, vision disturbances, inner-ear edema, and/or other sensory integration deficits.

Treatment of this particular population group has several challenges which include: 1) difficulty with early and specific injury assessment 2) the determination of appropriate return-to-duty measures 3) selection of effective individualized balance rehabilitation and treatment tools 4) Prolonged length of rehabilitation and uncertain measureable endpoints. The group is also highly variable in the nature and extent of balance deficits and cognitive and / or related psychological impairments. It appears that almost all subjects with mTBI show some susceptibility to vestibular or vestibular/ocular disorders.

After assessment of disequilibrium, rehabilitation is often a course of remedial physical therapy (PT). To affect change in mobility by standard physical therapy, sensory and motor systems are "habituated" through exercise, with hope of rehabilitating the system and "compensating" by instructing the patient to alter skill sets associated with a task. Compensation (without immediate sensory feedback) is problematic and prone to patient (and caregiver) interpretation and error, because it may not address the underlying problems and may not have long term therapeutic benefits. There is also a very limited pool of PTs who specialize in the treatment of neurological problems resulting from brain injuries. Individual vestibular rehabilitation treatment programs are designed by these specialist PTs who also monitor and participate in each patient's recovery. This approach is labor intensive, time consuming (up to 14 weeks of therapy is often needed) and some patients do not recover fully .

The overall objective of this research effort is to use novel combinations of multi-modal sensory guided feedback (especially tactile) and traditional vestibular rehabilitation to retrain military personnel suffering balance disorders as a result of mTBI. The investigators therapeutic goal is to test technology that will return the patient, in the shortest period of time, to a level of balance performance consistent with return to the community and/or military duty.

The sense of touch is intrinsically linked with the neuro-motor channel, both at the reflex and higher cognitive regions, which makes it uniquely tied to orientation and localization. Vibrotactile arrays are therefore intuitive and are an effective sensory feedback pathway.

Recent research has also demonstrated that tactile cueing yield significantly faster and more accurate performance than comparable spatial auditory cues. Further research has demonstrated this finding is relatively stable across a variety of body orientations, even when spatial translation is required and under physiological stress.

Over a Phase I SBIR and current Phase II effort, Engineering Acoustics Inc. has developed the Sensory Kinetics (SK) Balance System. In the SK system, patients move on a force platform (see Figure 1) while movement and posture data is interpreted by advanced software a mapped to a wearable vibrotactile belt array and visual display. Vibrotactile cueing provides continuous and instantaneous feedback to the patient that compliments their postural and mobility decisions. The investigators believe that vibrotactile feedback can greatly increase spatial awareness and consequently mobility. Further, the ability of the brain to re-organize and relearn functional movement activities provides an intriguing potential pathway for the retention of learned functional mobility strategies.Vibrotactile cueing involves short duration bursts of mechanical vibration from actuators, or tactors, that are mounted within a torso worn belt. The person's position is measured and calculated using a force plate sensor and camera sensors. The computerized system is then used as part of physical therapy balance training to improve the patient's balance and potentially reduce their risk of falling.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Traumatic Brain Injury
* Adults 18 years-75 years old
* Vestibular &/or balance deficit following mild/moderate TBI and confirmed by healthcare professional
* Subjects reporting head injury from exposure to a blast/concussion injury with one or more of the following symptoms: dizziness, vertigo, headache, migraine, oscillopsia, movement induced vertigo.
* Able to sit unaided for two minutes
* Able to stand independently with or without a cane, or with no more than moderate assistance from the physical therapist/researcher.

Exclusion Criteria:

* Multiple trauma
* Severe brain injury as defined above
* Pacemakers
* Weight greater than 250 lbs
* Mini Mental Status Exam score of less than 24 and/or Cognitive Log score of less than 25
* A diagnosis of:
* Peripheral neuropathy
* Severe neuromuscular diseases
* Severe Cardiovascular disease
* Associated high-level stroke or spinal cord injury
* Amputees

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Started | 16 | 15
Completed | 16 | 14
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (16.4) | 41.9 (9.6) | 42.2 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale
Description: The BBS is a 14-item objective measure designed to assess static balance and fall risk in adult populations and is a well-accepted measure in the stroke literature. The functional activities that are assessed include sitting and standing balance during transfers, altered base of support, reaching, turning, eyes open and closed. Each item is scored from 0 to 4 points. The maximum score is 56 points. A score from 0 to 20 represents balance impairment, 21 to 40 represents acceptable balance, and 41-56 represents good balance.
Time Frame: Pre-training,Midpoint Assessment (4 weeks), Post Training (8 weeks)
Measure: Mean (Standard Deviation); unit: Units on a continuous scale
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
Units on a continuous scale
  Pre training | 45 (10.94969558) | 44 (10.65338)
  Mid Training | 48 (10.83743512) | 47 (10.27212167)
  Post Training | 50 (8.932851355) | 47 (11.25649995)

2. Primary Outcome: Functional Gait Assessment (FGA)
Description: Assesses postural stability during walking tasks. This test is a modification of the Dynamic Gait Index (DGI) developed to improve reliability and decrease the ceiling effect.
  10-item test that comprises 7 of the 8 items from the original DGI Eliminated 1 item from original DGI, ambulation around obstacles Added 3 new items to the original DGI, including gait with narrow base of support, ambulating backwards, and gait with eyes closed were added Each item is scored on an ordinal scale from 0 - 3, with 0 = severe impairment
  1. = moderate impairment
  2. = mild impairment
  3. = normal ambulation Highest score = 30 Assessment may be performed with or without an assistive device
Time Frame: Pre-training, Mid-training assessment (4 weeks), Post-training (8 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
units on a scale
  Pre-training | 15.714 (6.51) | 17.125 (5.72)
  Mid-training assessment (4 weeks) | 18.929 (6.52) | 21.21 (6.65)
  Post-training (8 weeks) | 20.642 (6.52) | 23.36 (6.87)

3. Secondary Outcome: 10 Meter Walk Test
Description: assesses walking speed of short duration
Time Frame: Pre-training, mid training (4 weeks), post training (8 weeks)
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
m/s
  Pre-training | 0.873 (0.496) | 1.067 (0.532)
  Mid-training assessment (4 weeks) | 0.944 (0.617) | 1.236 (0.632)
  Post-training (8 weeks) | 1.021 (0.652) | 1.253 (0.749)

4. Secondary Outcome: Six Minute Walk Test
Description: Assesses distance walked over 6 minutes
Time Frame: Pre-training, mid training (4 weeks), post training (8 weeks)
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
Feet
  Pre-training | 1021.6 (544.1) | 1158.2 (490.5)
  Mid-training assessment (4 weeks) | 1075.4 (624.1) | 1271.1 (566.1)
  Post-training (8 weeks) | 1165.6 (662.1) | 1312.7 (627.5)

5. Secondary Outcome: Modified Clinical Test of Sensory Organization and Balance (mCTSlB) - Eyes Closed
Description: Clinical Test of Sensory Interaction and Balance (CTSIB): assesses balance under a variety of conditions including vision blocked and surface challenges.
  The patient performance is timed for 30 seconds. Test is terminated when a subject's arms or feet change position. If a patient in unable to maintain the position for 30 seconds they are provided with 2 additional attempts.
  The scores of the 3 trials are averages
Time Frame: Pre-training, mid training, post training
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
sec
  Pre-Training | 11.18375 (10.15539992) | 9.119280952 (7.06647348)
  Mid Training | 15.98062479 (12.19808074) | 16.99357119 (11.85259485)
  Post Training | 17.986458 (11.13131861) | 20.423095 (9.057258643)

6. Secondary Outcome: Modified Clinical Test of Sensory Organization and Balance (mCTSlB) - Eyes Open
Description: The mCTSIB provides the clinician with a means to quantify postural control under various sensory conditions.
  The patient performance is timed for 30 seconds. Test is terminated when a subject's arms or feet change position. If a patient in unable to maintain the position for 30 seconds they are provided with 2 additional attempts.
  The scores of the 3 trials are averages
Time Frame: Pre-training, mid training (4 weeks), post training (8 weeks)
Measure: Mean (Standard Deviation); unit: sec
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
sec
  Pre-training | 21.13041667 (10.59997686) | 21.13333333 (10.93591753)
  Mid Training | 27.039375 (10.71693518) | 25.715 (9.43461609)
  Post Training | 27.467271 (9.635670393) | 26.277143 (9.195793711)

7. Secondary Outcome: Activities Balance Confidence Scale (ABC)
Description: Subjective measure of confidence in performing various ambulatory activities without falling or experiencing a sense of unsteadiness.
  16-item self-report measure in which patients rate their balance confidence for performing activities. This stem is used to lead into each activity considered: "How confident are you that you will not lose your balance or become unsteady when you..." Items are rated on a rating scale that ranges from 0 - 100 Score of zero represents no confidence, a score of 100 represents complete confidence Overall score is calculated by adding item scores and then dividing by the total number of items
Time Frame: Pre-training, mid training, post training
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 16 | 14
units on a scale
  Pre-training | 60.1396875 (23.04021958) | 55.53035714 (23.85675041)
  Mid Training | 71.1828125 (21.01544763) | 60.11178571 (20.51856435)
  Post Training | 72.445313 (22.50808738) | 66.151786 (19.0398228)

8. Secondary Outcome: Dizziness Handicap Inventory
Description: A 25-item self-assessment inventory designed to evaluate the self-perceived handicapping effects imposed by dizziness. Participants complete the questionnaire only if they report dizziness.
  Self-report questionnaire Quantifies the impact of dizziness on daily life by measuring self-perceived handicap Three domains: functional (9 questions, 36 points), emotional (9 questions, 36 points), and physical (7 questions, 28 points) Maximum score of 100 (28 points for physical, 36 points for emotional and 36 points for functional) to Minimum score of 0. The higher the score, the greater the perceived handicap due to dizziness Item scores are summed Answers are graded 0 (no), 2 (sometimes) and 4 (yes)
Time Frame: Pre-training, mid training, post training
Population: This data includes the participants in this study that self reported yes to dizziness. If they answered no to dizziness they did not have the scale administered to them.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Number analyzed (Participants) | 10 | 4
Units on a scale
  Pre-training | 40.6 (26.87) | 40.5 (10.88)
  Mid Training | 37.0 (28.41) | 38.5 (11.47)
  Post Training | 32.6 (25.58) | 26.0 (9.09)

ADVERSE EVENTS:
Description: 0% Indicates that no adverse events were encountered during the study.
Arm/Group | Sensory Kinectics Balance System | Traditional Vestibular Rehabilitation
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No